CLINICAL TRIAL: NCT06190561
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE-DOSE, PARALLEL DESIGN, STUDY TO EVALUATE PHARMACOKINETIC COMPARABILITY OF TWO PF-07940367 FILM-COATED TABLET FORMULATIONS ADMINISTERED AS 150 MG UNDER FASTED CONDITIONS IN HEALTHY PARTICIPANTS
Brief Title: A Study to Learn How Different Products of the Study Medicine Called PF-07940367 Are Taken up Into the Blood in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C5351008; GBT BEFE (adult formulation) (Other: Alias Study Number)
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: PF-07940367 Product II (Experimental): tablet by mouth
  Interventions: Drug: PF-07940367
- Treatment B: PF-07940367 Product I (Experimental): tablet by mouth
  Interventions: Drug: PF-07940367

INTERVENTIONS:
Drug: PF-07940367 — Participants to receive a single dose of PF-07940367 product II 150 mg by mouth
  Arms: Treatment A: PF-07940367 Product II
Drug: PF-07940367 — Participants to receive a single dose of PF-07940367 product I 150 mg by mouth
  Arms: Treatment B: PF-07940367 Product I

SUMMARY:
The purpose of this study is to compare two finished products of PF-07940367 in terms of the uptake into the blood stream.

This study is seeking participants who are:

- Healthy male or female participants aged 18 years or older.

All participants in this study will receive PF-07940367 once by mouth. The participants may receive different tablets by mouth for PF-07940367.

The study will compare experiences of people receiving two different products of PF-07940367. This will help understand how much PF-07940367 is taken up into the blood for each product given.

Participants will take part in the study for about 112 days. During this time, participants will have to stay onsite for 5 days. There will be up to 2 additional onsite study visits and 3 remote (telephone call) study visits.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* BMI of 16-32 kg/m2; and a total body weight >50 kg (110 lb).
* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations and other study procedures.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in the protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis A, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis B surface antigen (HCVAb). Hepatitis B vaccination is allowed.
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription drug, dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.
* A positive urine drug test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Area under the whole blood concentration versus time curve (AUC) from time zero (pre-dose) to 336 hours (AUC336) of PF-07940367 dose to evaluate pharmacokinetic comparability of two PF-07940367 products | 0 hours (pre-dose) to 336 hours post-PF-07940367 dose

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) | From baseline up to 56 days after PF-07940367 dose
Number of Participants With Clinically Significant Laboratory Abnormalities | From baseline up to 336 hours after PF-07940367 dose
Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings | From baseline up to 96 hours after PF-07940367 dose
Number of Participants With Clinically Significant Vital Signs | From baseline up to 336 hours after PF-07940367 dose
Maximum Observed Whole Blood Concentration (Cmax) of PF-07940367 for two PF-07940367 products | 0 hours (pre-dose) to 336 hours post-PF-07940367 dose
Area under the whole blood concentration versus time curve (AUC) from time zero (pre-dose) to the last quantifiable concentration (AUClast) of PF-07940367 for two PF-07940367 products | 0 hours (pre-dose) to 336 hours post-PF-07940367 dose
Time to Maximum Observed Whole Blood Concentration (Tmax) of PF-07940367 for two PF-07940367 products | 0 hours (pre-dose) to 336 hours post-PF-07940367 dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5351008